CLINICAL TRIAL: NCT02873091
Title: Comparison of Programmed Intermittent Epidural Bolus With Continuous Epidural Infusion for Labor Epidural Analgesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Maternity and Child Health Care Hospital (Other)
Responsible Party: Principal Investigator, Caijuan Li, Nanjing Maternity and Child Health Care Hospital, Nanjing Maternity and Child Health Care Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NJFY2016002
Record Dates: First submitted 2016-08-11; First posted 2016-08-19 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-12

CONDITIONS: Labor Analgesia
MeSH Terms: interventions — Analgesia, Epidural; Ropivacaine; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CEI (Active Comparator): Initial loading dose:10 ml (0.125% ropivacaine with 0.4 μg/ml sufentanil) Epidural infusion with maintain dose: 0.08% ropivacaine with 0.4 μg/ml sufentanil. The basal infusion of CEI: 10 ml/h, beginning immediately after the initial dose
  Interventions: Procedure: Epidural analgesia; Procedure: Continuous epidural infusion; Drug: ropivacaine; Drug: sufentanil
- PIEB 1 (Active Comparator): Initial loading dose:10 ml (0.125% ropivacaine with 0.4 μg/ml sufentanil) Epidural infusion with maintain dose: 0.08% ropivacaine with 0.4 μg/ml sufentanil.The basal infusion of PIEB1: 5 ml per 30 min, beginning 30 min after the initial dose
  Interventions: Procedure: Epidural analgesia; Procedure: Intermittent epidural bolus; Drug: ropivacaine; Drug: sufentanil
- PIEB 2 (Active Comparator): Initial loading dose:10 ml (0.125% ropivacaine with 0.4 μg/ml sufentanil) Epidural infusion with maintain dose: 0.08% ropivacaine with 0.4 μg/ml sufentanil. The basal infusion of PIEB2: 10 ml per 60 min, beginning 60 min after the initial dose
  Interventions: Procedure: Epidural analgesia; Procedure: Intermittent epidural bolus; Drug: ropivacaine; Drug: sufentanil

INTERVENTIONS:
Procedure: Epidural analgesia
Procedure: Continuous epidural infusion
  Arms: CEI
Procedure: Intermittent epidural bolus
  Arms: PIEB 1; PIEB 2
Drug: ropivacaine
Drug: sufentanil

SUMMARY:
Sixteen million babies were born in 2010, approximately half were by cesarean. Labor analgesia should be the first choice for these parturients based on the consideration of security and humanization. However this labor analgesia rate is quite low in China (<5%) while in western country, this rate is up to 60%. Programmed intermittent epidural bolus (PIEB) is the latest technique for labor analgesia which has less neurotoxicity theoretically compared with Continuous Epidural Infusion(CEI) with Patient controlled epidural analgesia (PCEA) which is used most commonly. In that study, they reported less total local anesthetic consumption, fewer manual bolus doses and greater patient satisfaction with the PIEB technique. In China, multiple factors contribute to the reasons of low labor analgesia rate. From the patient's point of view, worrying about unsatisfied analgesia, and not adapted to the symptoms of motor block, such as inability to move their legs distressing, both are important reasons of refusing labor analgesia and preferring to cesarean delivery. Therefore, in this clinical trial, we plan to find a safer and more effective regimen for labor analgesia in Chineseparturients. This clinical trial is designed to prove PIEB used Ropivacaine is safer and more effective than CEI for labor analgesia in Chinese parturients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who agree to join this study
* Age: 22y-40y
* American Society of Anesthesiologists (ASA) physical status 1 or 2
* Gestation : 37-41 weeks
* Primipara
* Singleton fetus and head presentation
* In early labor: cervical dilation for 1-3cm
* Requesting labor epidural analgesia

Exclusion Criteria:

* Contraindication for epidural analgesia
* Height less than 150 cm or more than 170 cm
* Morbid obesity (BMI more than 35)
* High-risk pregnancy:(gestational diabetes mellitus, gestational hypertension, placenta previa, placental abruption, preeclampsia)
* Received parenteral opioids
* Unable to perform motor block evaluation tests

Ages: 22 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 186 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-05 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Maternal visual analogue scale (VAS) | At time of initiation of analgesia and hourly thereafter until 1 hours postpartum (approximately 10 hours)
  a visual analog scale (VAS) with a 10 cm vertical score ranged from "no pain" to "worst possible pain"

SECONDARY OUTCOMES:
Maternal modified Bromage scale | At time of initiation of analgesia and hourly thereafter until 2 hours postpartum (approximately 10 hours)
Subject's Satisfaction with labor epidural analgesia | At the time after childbirth
Total ropivacaine and sufentanil consumption | At two hours postpartum
Proportion of parturients requiring additional PCEA boluses | At two hours postpartum
Rate of "very satisfied"and/or "satisfied",Proportion of subjects who has experienced Visual analog scale (VAS) score for pain more than 3 scale | At two hours postpartum
Maternal heart rate | At time of initiation of analgesia and hourly thereafter until 4 hours postpartum (approximately 12 hours)
Rates of cesarean delivery and instrument-assisted delivery | At time of placental delivery
Duration of analgesia | Initiation of analgesia to 2 h postpartum (approximately 10 hours)
Durations of labor stages | From the beginning of regular contraction of uterus to the end of the labor (approximately 12 hours)
Use of oxytocin after analgesia | At twenty-four hours postpartum
Incidence of maternal side effects | Initiation of analgesia to 2 hour postpartum (approximately 10 hours)
Neonatal Apgar scale | At the first and fifth minutes after baby was born
Fetal heart rate | From initiation of analgesia to delivery (approximately 8 hours)
Neonatal weight | At delivery
Mean number of PCEA | At two hours postpartum
Maternal respiratory rate | At time of initiation of analgesia and hourly thereafter until 4 hours postpartum (approximately 12 hours)
Maternal blood pressure | At time of initiation of analgesia and hourly thereafter until 4 hours postpartum (approximately 12 hours)

CONTACTS AND LOCATIONS:
Locations (1):
- Obstetrics and Gynecology Hospital Affiliated to Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No